CLINICAL TRIAL: NCT00898430
Title: Biomarkers of Survival in HNSCC
Brief Title: Biomarkers in Predicting Response to Treatment in Patients With Newly Diagnosed Stage III or Stage IV Head and Neck Cancer Treated With Carboplatin, Paclitaxel, and Radiation Therapy
Status: Terminated | Type: Observational
Why Stopped: Study closed prematurely upon PI's departure
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC HN 0392; P30CA068485 (NIH); VU-VICC-HN-0392; VU-VICC-030933
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; untreated metastatic squamous neck cancer with occult primary; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; salivary gland squamous cell carcinoma; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Oligonucleotide Array Sequence Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Head and neck squamous cell carcinoma patients (HNSCC)
  Interventions: Genetic: DNA Microarray analysis; Genetic: MALDI-TOF mass spectrometry; Genetic: DNA microarray and MALDI-TOF mass spectrometry

INTERVENTIONS:
Genetic: DNA Microarray analysis — Tumors will be assayed on Affymetrix Human Genome U133 GeneChip
Genetic: MALDI-TOF mass spectrometry — Supervised analysis techniques will be employed to identify patterns of protein peaks useful for treatment response and survival prediction. Hierarchical clustering analyses will be used to visualize data.
Genetic: DNA microarray and MALDI-TOF mass spectrometry — Tumors from the specific Aim 1/2 and from preliminary data, previously analyzed, will be examined for HPV 16 infection.

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at biomarkers in predicting response to treatment in patients with newly diagnosed stage III or stage IV head and neck cancer treated with carboplatin, paclitaxel, and radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if gene expression patterns that correlate with treatment response and survival can be identified using DNA microarrays in patients with newly diagnosed head and neck squamous cell carcinoma (HNSCC) treated with carboplatin, paclitaxel, and radiotherapy.
* Determine if protein expression patterns that correlate with treatment response and survival in HNSCC can be identified using matrix-assisted laser desorption ionization-time-of-flight mass spectrometry (MALDI-TOFMS).
* Determine if the molecular signature of human papilloma virus-16 infection can be determined using DNA microarray and MALDI-TOFMS and correlate with gene and protein expression, treatment response, and survival.

OUTLINE: Tumor tissue samples are analyzed by DNA microarray analysis and validated by quantitative reverse transcription-polymerase chain reaction (PCR). Protein and gene expression patterns are analyzed by laser desorption ionization-time-of-flight mass spectrometry, high performance liquid chromatography, liquid chromatography-tandem mass spectrometry, and PCR. Samples are also analyzed by tissue microarray and immunohistochemistry.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed head and neck squamous cell carcinoma

  * Stage III-IV disease
* Scheduled for pan-endoscopy
* Tumor tissue available from patients treated with carboplatin, paclitaxel, and radiotherapy on protocol VU-VICC-HN-0356

PATIENT CHARACTERISTICS:

* Able to speak English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Head and Neck cancer patients who are uniformly treated with concurrent carboplatin/paclitaxel and radiation.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2003-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Survival | at expiration of last patient enrolled

SECONDARY OUTCOMES:
Treatment response | upon patient tissue collection

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee